CLINICAL TRIAL: NCT01567449
Title: Risk Factors in Predicting Spontaneous Intracranial Aneurysm Rebleeding During Hospitalization
Brief Title: Risk Factors for Aneurysm Rebleeding
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Qingsong Lin, Junior Doctor of Neurosurgery,Principal Investigator,Clinical Doctor, Fujian Medical University
Other Study IDs: 110011
Record Dates: First submitted 2012-03-25; First posted 2012-03-30 (Estimated); Last update posted 2012-03-30 (Estimated); Status verified 2012-03

CONDITIONS: Subarachnoid Hemorrhage, Aneurysmal
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- the case group: The case group referred to SAH patients with aneurysm rebleeding
- the control group: the control group referred to SAH patients not with aneurysm rebleeding

SUMMARY:
The purpose of this study is to examine the risk factors for aneurysm rebleeding.

DETAILED DESCRIPTION:
To investigate risk factors for spontaneous aneurysm rebleeding during hospitalization and to reach conclusions if any,of clinical signs for predicting rebleeding.

ELIGIBILITY:
Inclusion Criteria:

* Individual whose clinical course was clear enough to be traced back and whose conservative treatment duration was shorter than 6 weeks was included

Exclusion Criteria:

* Rebleeding patients with certain inducing factors such as:

  * severe emotional episode,
  * severe coughing,
  * constipation,
  * excessive activities, or
  * with coagulation disorder,or
  * with other intracranial vascular malformations,such as:

    * moyamoya disease,
    * arteriovenous malformation were excluded.
* Also patients who rebled while angiography were excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A total of 66 SAH patients were enrolled in this study
Sampling Method: Non-Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2011-09; Primary Completion 2012-03 (Actual); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
Aneurysm rebleeding | up to 7 months

CONTACTS AND LOCATIONS:
Overall Officials: Dezhi kang, professor, Study Director — First Affiliated Hospital of Fujian Medical University
Locations (1):
- First Affiliated Hospital,Fujian Medical University, Fuzhou, Fujian, China